CLINICAL TRIAL: NCT02617069
Title: Botulinum Toxin Injection Into Epicardial Fat Pads to Prevent Atrial Fibrillation in Patients Undergoing Cardiac Surgery: Randomized Study
Brief Title: Botulinum Toxin Injection Into Epicardial Fat Pads to Prevent Atrial Fibrillation in Patients Undergoing Cardiac Surgery
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NTPAF-01
Record Dates: First submitted 2015-11-25; First posted 2015-11-30 (Estimated); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; botulinum toxin
MeSH Terms: conditions — Atrial Fibrillation | interventions — Botulinum Toxins; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Cardiac surgery+botulinum toxin) (Experimental): All patients underwent conventional cardiac surgery. After the main stage of the surgery botulinum toxin (50 U/1 mL) was injected into the entire four visible area of the major epicardial fat pads. First epicardial left atrial fat pad is located anterior to the right superior pulmonary vein and corresponding to the anterior right ganglionated plexi (GP); second epicardial fat pad is located inferoposterior to the right inferior pulmonary vein and corresponding to the inferior right GP; third fat pad is located anterior to the left superior pulmonary vein (PV) and left inferior PV (between the PVs and left atrial appendage (LAA), corresponding to the Marshall tract GP and superior left GP; forth fat pad located inferiorly to the left inferior PV and extends posteriorly and corresponding to the inferior left GP
  Interventions: Biological: botulinum toxin injection; Device: Implantable loop recorder
- Group 2 (Cardiac surgery+placebo) (Active Comparator): All patients underwent conventional cardiac surgery. After the main stage of the surgery 0.9% normal saline (1 mL at each fat pad) was injected into the entire four visible area of the major epicardial fat pads. First epicardial left atrial fat pad is located anterior to the right superior pulmonary vein and corresponding to the anterior right GP; second epicardial fat pad is located inferoposterior to the right inferior pulmonary vein and corresponding to the inferior right GP; third fat pad is located anterior to the left superior PV and left inferior PV (between the PVs and LAA), corresponding to the Marshall tract GP and superior left GP; forth fat pad located inferiorly to the left inferior PV and extends posteriorly and corresponding to the inferior left GP
  Interventions: Biological: 0.9% normal saline injection; Device: Implantable loop recorder

INTERVENTIONS:
Biological: botulinum toxin injection
  Arms: Group 1 (Cardiac surgery+botulinum toxin)
Biological: 0.9% normal saline injection
  Arms: Group 2 (Cardiac surgery+placebo)
Device: Implantable loop recorder

SUMMARY:
The aim of this prospective randomized double-blind study was to compare the efficacy of botulinum toxin injection in epicardial fat pads for preventing recurrences (in early postoperative period) of atrial tachyarrhythmia in patients undergoing cardiac surgery.

ELIGIBILITY:
Key inclusion Criteria:

* Indication for cardiac surgery (e.g. coronary artery bypass grafting, valve repair/replacement) according to the American College of Cardiology/American Heart Association (ACC/AHA) guidelines for cardiac surgery

Key exclusion Criteria:

* Planned maze procedure or pulmonary vein isolation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-03 (Actual); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Recurrence of >30 s of any atrial tachyarrhythmia, including atrial fibrillation (AF) and atrial flutter/tachycardia, after cardiac surgery procedure with no antiarrhythmic drug. | 1 month

SECONDARY OUTCOMES:
Recurrence of >30 s of any atrial tachyarrhythmia, including AF and atrial flutter/tachycardia, after cardiac surgery procedure with no antiarrhythmic drug. | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- State Research Institute of CIrculation Pathology Novosibirsk, Russian Federation, Novosibirsk, Russia